CLINICAL TRIAL: NCT02720783
Title: A Phase I Study of a Novel Antimycotic Vaginal Pessary Formulation (Econazole Nitrate 150 mg + Benzydamine HCl 6 mg) Administered Once Daily for 3 Days to Healthy Women
Brief Title: Tolerability and Pharmacokinetic Study of Econazole Nitrate Plus Benzydamine HCl Vaginal Pessary
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 030(4C)HO15323; CRO-PK-15-302 (Other: CROSS Research S.A., Phase I Unit)
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Healthy Women
Keywords: Pharmacokinetics; Econazole nitrate 150mg; Benzydamine HCl 6mg; Vaginal pessary; Tolerability
MeSH Terms: interventions — Econazole; Benzydamine; Suppositories

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Econazole nitrate 150 mg plus Benzydamine HCl 6 mg (Experimental): One vaginal pessary (2.7 g) of Econazole nitrate 150 mg plus Benzydamine HCl 6 mg, once daily, for 3 consecutive days
  Interventions: Drug: Econazole nitrate 150 mg plus Benzydamine HCl 6 mg vaginal pessary
- Placebo plus Econazole nitrate 150 mg (Active Comparator): One vaginal pessary (2,7 g) of Placebo plus Econazole nitrate 150 mg, once daily, for 3 consecutive days
  Interventions: Drug: Placebo plus Econazole nitrate 150 mg vaginal pessary
- Placebo plus Benzydamine HCl 6 mg (Active Comparator): One vaginal pessary (2,7 g) of Placebo plus Benzydamine HCl 6 mg, once daily, for 3 consecutive days
  Interventions: Drug: Placebo plus Benzydamine HCl 6 mg vaginal pessary
- Placebo (Placebo Comparator): One vaginal pessary (2.7 g) of Placebo, once daily, for 3 consecutive days
  Interventions: Drug: Placebo vaginal pessary

INTERVENTIONS:
Drug: Econazole nitrate 150 mg plus Benzydamine HCl 6 mg vaginal pessary — Econazole nitrate 150 mg plus Benzydamine HCl 6 mg vaginal pessary
  Arms: Econazole nitrate 150 mg plus Benzydamine HCl 6 mg
Drug: Placebo plus Econazole nitrate 150 mg vaginal pessary
  Arms: Placebo plus Econazole nitrate 150 mg
Drug: Placebo plus Benzydamine HCl 6 mg vaginal pessary
  Arms: Placebo plus Benzydamine HCl 6 mg
Drug: Placebo vaginal pessary
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the local tolerability of the new Econazole/Benzydamine pessary, in comparison with Econazole and Benzydamine stand-alone products and placebo. Pharmacokinetics of the study products after single and multiple applications o.d. for 3 days, overall local and general tolerability, safety and comfort of use will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study.
2. Sex and age: healthy women, aged 18-55 years old inclusive.
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive.
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest (sitting position).
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study.
6. Sexual abstinence: agreement to sexual abstinence during the study.
7. Contraception and fertility: women of child-bearing potential, even if sexually abstinent during the study as required by the study inclusion criteria, must be using at least one reliable method of contraception, as follows:

   1. hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit;
   2. a non-hormonal intrauterine device [IUD] for at least 2 months before the screening visit;
   3. a male sexual partner who agrees to use a male condom;
   4. a vasectomised sexual partner. Female participants of non-child-bearing potential will be admitted. For all female subjects, pregnancy test result must be negative at screening and on day 1.
8. PAP test: negative PAP test result (i.e. normal PAP test result without atypical cells) at screening.

Exclusion Criteria:

1. ECG (12-leads, supine position): clinically significant abnormalities.
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study as judged by the Investigator.
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness.
4. Allergies: ascertained or presumptive hypersensitivity (including allergies) to the active ingredients (econazole nitrate and/or benzydamine HCl) and/or formulations' excipients or related drugs, e.g. other azoles; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study.
5. Diseases: relevant history of renal, hepatic, gastrointestinal, genitourinary, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study or affect the subject's safety.
6. Genitourinary diseases: presence of any specific genitourinary symptoms detected at visit 2 with the relevant questionnaire (genitourinary symptoms questionnaire).
7. Infection history: history of bacterial urinary tract or bacterial or fungal vaginal infections for 3 weeks before the screening visit.
8. Systemic and/or local infections: bacterial or fungal infections that may interfere with the aim of the study or affect the subject's safety. If the results of the microbiological analyses concerning Ureaplasma/Mycoplasma and Actinomyces are positive, the subject can be enrolled only if asymptomatic and without any clinical evidence (gynaecological visit, PAP test and vaginal pH measurement) of vaginal infections.
9. Gynaecological findings: clinically significant abnormal findings at the gynaecological visit performed by the study Gynaecologist.
10. Mucosa conditions: altered mucosa conditions affecting the site of insertion (e.g. open lesions or other).
11. Habits: use of vaginal detergents, soaps and washes that, in the Investigator's opinion, may have an influence on vaginal pH and/or change the vaginal flora.
12. Medications: any medication (topical or systemic), including over the counter, herbal medication, topical drugs on the application area, and anticoagulants, such as warfarin, acenocoumarol and rivaroxaban, for 2 weeks before the start of the study. Hormonal contraceptives and hormonal replacement therapies are allowed. Paracetamol will be allowed as a counter-measure for adverse events, on a case by case basis, if deemed appropriate by the Investigator.
13. Investigative drug studies: participation in the evaluation of any drug for 3 months before this study, calculated from the first day of the month following the last visit of a previous study and the first day of the present study (date of the informed consent signature).
14. Blood donation: blood donations for 3 months before this study.
15. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (> 1 drink/day, defined according to USDA Dietary Guidelines 2010), tobacco (≥ 10 cigarettes/day) or caffeine (> 5 cups coffee/tea/day) abuse.
16. Diet: Abnormal diets (< 1600 or > 3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians.
17. Pregnancy: positive or missing pregnancy test at screening or day 1, pregnant or lactating women or females of child-bearing potential not following adequate contraceptive procedures.
18. Non-compliance: subjects suspected to have a high potential for non-compliance to the study procedures according to the Investigator's judgement, including non-compliance to sexual abstinence during the study.
19. Drug test (cocaine, amphetamine, methamphetamine, cannabinoids, opiates and ecstasy): positive result at the drug test at screening.
20. Alcohol test: positive alcohol breath test at day 1.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Local Adverse Drug Reactions (ADRs) | Up to 7 days after administration
  Occurence of local ADRs reported by the subjects as 1-3 scores for pruritus, burning sensation, pain, stinging and dryness; occurrence of all the other local Adverse Events (AEs) referred by the subjects; occurrence of all the local ADRs revealed by the Investigator/ Gynaecologist

SECONDARY OUTCOMES:
Econazole (free base), benzydamine (free base) and benzydamine N-oxide (free base) plasma concentrations | At pre-dose (0), 1, 2, 3, 4, 6, 8, 12, 24 hours after the first (day 1) and the last dose (day 3)
Area under the plasma concentration versus time curve [AUC(0-t)] of econazole (free base), benzydamine (free base) and benzydamine N-oxide (free base) | At pre-dose (0), 1, 2, 3, 4, 6, 8, 12, 24 hours after the first (day 1) and the last dose (day 3)
Overall local tolerability assessment scale | At final visit (from day 5 to day 8)
Occurrence of all AEs and ADRs | 5-8 days
Change from screening in laboratory parameters | From screening (from day -21 to day -7) at final visit (from day 5 to day 8)
Questionnaire for the comfort of use | At final visit (from day 5 to day 8)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A. Phase I Unit
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Stefano AFD, Radicioni MM, Vaccani A, Caccia G, Focanti F, Salvatori E, Pelacchi F, Picollo R, Rosignoli MT, Olivieri S, Bovi G, Comandini A. Phase I Study in Healthy Women of a Novel Antimycotic Vaginal Ovule Combining Econazole and Benzydamine. Infect Dis Obstet Gynecol. 2020 May 2;2020:7201840. doi: 10.1155/2020/7201840. eCollection 2020. PMID 32410819